CLINICAL TRIAL: NCT05977790
Title: Determinant of Fetal Growth Retardation After Sleeve Gastrectomy: Involvement of Ghrelin
Acronym: FG-SLEEVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220714
Record Dates: First submitted 2023-06-19; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: In Utero Growth Retardation; Sleeve Gastrectomy; Bariatric Surgery Status Complicating Pregnancy
Keywords: sleeve gastrectomy; ghrelin
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to determine, in pregnant women who have undergone sleeve gastrectomy (SG), whether ghrelin changes could be involved in in utero growth restriction (IUGR) and whether therefore a correlation between maternal ghrelin levels and birth weight is observed.

DETAILED DESCRIPTION:
Bariatric surgery (BS) has developed rapidly in recent years and the candidates are predominantly women of childbearing age. A negative impact on fetal growth (FG), has been described after BS whose mechanisms are not elucidated. The sleeve gastrectomy (SG), the most commonly practiced BS technique, is supposed to induce fewer nutritional deficiencies than gastric bypass. This is why it seems to be the technique of choice for young women, although the lack of hindsight does not allow recommendations to be made.

However, latest work showed that birth weight (BW) was affected as much after SG as after RYGB (Roux-en-Y Gastric Bypass), with 50% of BW Z-score <0 and 19% of small newborns for gestational age. In addition, only weight gain during pregnancy and maternal protein status were related to BW, but these parameters explained only 16% and 8% of the variance of the BW Z-score, respectively, suggesting that other factors are therefore involved.

Sleeve gastrectomy induces the loss of the majority of gastric cells secreting ghrelin, an orexigenic hormone involved in the regulation of appetite but also in the pituitary secretion of growth hormone, which could influence fetal growth, as shown in a model of pregnant rats. However, no studies have evaluated the link between maternal ghrelin and pregnancy outcome in women undergoing bariatric surgery.

The study population will include pregnant women who have undergone bariatric surgery such as sleeve gastrectomy (which is currently the most frequently performed technique) before pregnancy, coming to consult between the 3rd and 6th month of pregnancy (2nd trimester) for a nutritional check-up in a day hospital.

ELIGIBILITY:
Inclusion Criteria:

* Woman previously operated of sleeve gastrectomy
* Pregnant from 3 to 6 months
* Having a mono-fetal pregnancy
* Coming to consult in day hospital for a nutritional assessment

Exclusion Criteria:

* Twin pregnancy
* Identified cause of IUGR apart from those related to sleeve gastrectomy
* Woman who has undergone another bariatric surgery technique
* Lack of individual information and collection of the consent form
* Problems of understanding
* Lack of affiliation to a social security scheme or state medical aid
* Patient benefiting from a legal protection measure (with guardians or curators)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Study Population: The study population will include pregnant women who have undergone bariatric surgery such as sleeve gastrectomy before pregnancy, coming to consult between the 3rd and 6th month of pregnancy (2nd trimester) for a nutritional check-up in a day hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Correlation between ghrelin levels and birth weight of children born to mothers who had a sleeve gastrectomy | 18 months
  Fasting blood ghrelin level measured in plasma by radioimmunoassay technique in the second trimester of pregnancy. The dosages will be carried out deferred after freezing at -80 ° C in a laboratory, in order to be able to dose all the samples at the same time and limit the variability of the results.

SECONDARY OUTCOMES:
Nutritional factors that may influence birth weight after sleeve gastrectomy | 18 months
  These parameters will be collected between the 3rd and 6th month of pregnancy and childbirth.
  Parameters collected : parity, tobacco, alcohol, current treatment, vitamin supplementation, weight and BMI before sleeve, weight loss after sleeve, weight gain during the visit, caloric intake during the visit, number and type of nutritional deficiencies, total weight gain during pregnancy.
Obstetric factors that may influence birth weight after sleeve gastrectomy | 18 months
  These parameters will be collected between the 3rd and 6th month of pregnancy and childbirth.
  Parameters collected : term at time of analysis, time since sleeve, term of pregnancy at birth, sex of child, PN Z-score, complications of pregnancy or birth
Nutritional factors that may interact with the effect of ghrelin | 18 months
  These parameters will be collected between the 3rd and 6th month of pregnancy and childbirth.
  Parameters collected : parity, tobacco, alcohol, current treatment, vitamin supplementation, weight and BMI before sleeve, weight loss after sleeve, weight gain during the visit, caloric intake during the visit, number and type of nutritional deficiencies, total weight gain during pregnancy.
Obstetric factors that may interact with the effect of ghrelin | 18 months
  These parameters will be collected between the 3rd and 6th month of pregnancy and childbirth.
  Parameters collected : term at time of analysis, time since sleeve, term of pregnancy at birth, sex of child, PN Z-score, complications of pregnancy or birth

CONTACTS AND LOCATIONS:
Overall Officials: Séverine Ledoux, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Louis Mourier, Colombes, France

IPD SHARING:
Plan to Share IPD: No